CLINICAL TRIAL: NCT01845870
Title: Study Whether Serum 1,25-dihydroxyvitamin D Levels Could be an Indicator for Dysfunction of Renal Tubules
Brief Title: Serum 1,25-dihydroxyvitamin D Levels in Type 2 Diabetes Mellitus Patients With Different Levels of Albuminuria
Acronym: DM
Status: Completed | Type: Observational
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Fei Guo, chief physician, Tianjin Medical University General Hospital
Other Study IDs: TIJMUGHE
Record Dates: First submitted 2013-04-26; First posted 2013-05-03 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-04

CONDITIONS: Type 2 Diabetes Mellitus With Diabetic Nephropathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Blood samples were collected after an overnight fast to evaluate glycosylated hemoglobin A1c（HbA1c）, hemoglobin (Hb), serum albumin (ALB), serum creatinine (SCR), serum urea nitrogen (BUN), uric acid (UA), serum calcium (Ca), serum phosphate (P), serum alanine transferase (ALT), serum aspartate aminotransferase (AST), serum alkaline phosphatase (ALP), serum 25-hydroxyvitamin D and 1,25-dihydroxyvitamin D. Urine albumin, calcium and phosphate of 24 hour were also evaluated.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- urinary albumin >300mg/24h: none extra intervention was given by the investigator
- urinary albumin <30mg/24h: none extra intervention was given by the investigator
- urinary albumin 30 to 300mg/24h: none extra intervention was given by the investigator

SUMMARY:
Diabetic nephropathy(DN)is a major microvascular complication of diabetes.Renal injury may be presented with the characteristics of albuminuria, and its main pathological change is glomerular sclerosis. However, both glomerular lesions such as glomerulosclerosis, glomerular basement membrane thickness and tubulointerstitial fibrosis have been found in both type 1 and type 2 diabetic patients with normal urinary albumin excretion rate, moreover the tubular injury may be the primary pathological change in diabetic renal injury not only the secondary change brought on by glomerular injury. Thus, if overt urinary albumin exists in T2DM patients, the tubular injury may be severe already. An index which is predominant, sensitive and convenient to be measured should be purposed.It is predicted that insufficient renal 1-alpha hydroxylase may play a critical role in diabetic nephropathy. Then the investigators present the presumption that the activity of renal 1-alpha hydroxylase could reflect the degrees of tubulointerstitial injury, using serum 1,25-dihydroxyvitamin D level as an index.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years, DM duration >1 year, all of the patients were predialysis

Exclusion Criteria:

* history of liver or kidney disease, malignancy, current pregnancy, extensive dermatologic disease, evidence of metabolic bone disease and hyper-/hypo- thyroidism that would affect mineral metabolism. Patients who were taking native or active vitamin D, steroids, phosphate binders, or medications that affect vitamin D metabolism were also excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with T2DM were recruited from the general hospital of Tianjin Medical University in China .
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2012-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
determination of urinary albumin | 8 weeks
  Urinary albumin of 24h were measured by Scientific Management of HITACHI 7600-020 Biochemical Analyzer.

SECONDARY OUTCOMES:
determination of serum vitamin D metabolites | 8 weeks
  Serum vitamin D metabolites were detected by VITROS ECI systerm through a ELISA methods.

CONTACTS AND LOCATIONS:
Overall Officials: Chenlin Dai, MD, Study Director — Tianjin Medical University General Hospital
Locations (1):
- General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality, China